CLINICAL TRIAL: NCT07392970
Title: A Pilot Clinical Trial of Motixafortide for Measurable Residual Disease (MRD) Sensitization in Acute Myeloid Leukemia (AML)
Brief Title: Motixafortide for MRD Sensitization in AML
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Gamida Cell ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 26-x009
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Measurable Residual Disease
Keywords: AML; MRD; NGS; PCR
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Motixafortide Injection (Experimental): Consenting and eligible patients will bone marrow and peripheral blood testing assessments along with measurable residual disease (MRD) assays. Following completion of assessments, patients will receive a single injection of Motixafortide. The following day, 10-14 hours after the injection, patients will repeat the peripheral blood testing for MRD tests. Investigators will follow up with patients every 4 months for 18 months after study treatment.
  Interventions: Drug: Motixafortide

INTERVENTIONS:
Drug: Motixafortide — Motixafortide is a CXCR4 inhibitor for the mobilization of hematopoietic stem progenitor cells (HSPCs) in patients undergoing autologous stem cell transplantation. It is provided as a single subcutaneous injection.
  Other Names: Aphexda

SUMMARY:
This is a pilot phase I study evaluating the effect of motixafortide on determination of measurable residual disease (MRD) level in patients with acute myeloid leukemia (AML) who have completed induction treatment. Consenting and eligible patients will undergo standard of care (SOC) bone marrow and peripheral blood assessments with SOC MRD assays, followed by a single injection of motixafortide. Ten to 14 hours after injection, the patient will undergo peripheral blood collection for the same applicable MRD tests

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute myeloid leukemia (AML), excluding APL, treated with 1-2 cycles of front-line chemotherapy.
* Achieved CBC parameters compatible with complete remission (CR), complete remission with incomplete hematologic recovery (CRi), or complete remission with partial hematologic recovery (CRh) as defined by ELN 2022. This must be done within 5 days prior to study enrollment.
* Planning to undergo a standard of care blood draw and bone marrow assessment with SOC MRD assays, including morphology, flow cytometry for MRD, NGS panels for MRD, and PCR tests for MRD as applicable.
* At least 18 years of age.
* ECOG performance status ≤ 2
* Life expectancy > 3 months.
* Adequate organ function as defined below:

  * Total bilirubin ≤ 2.0 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 5.0 x IULN
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Evidence of more than 5% blasts in in the peripheral blood by manual differential within 5 days prior to study enrollment.
* Prior history of allogeneic stem cell transplant.
* Prior or concurrent malignancy whose natural history has the potential to interfere with the safety or efficacy assessment of the investigational regimen. Patients with prior or concurrent malignancy that does NOT meet that definition are eligible for this trial
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to motixafortide.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia. Patients with a known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Function Classification; to be eligible for this trial, patients should be a class 2B or better.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* HIV-infected if not on effective anti-retroviral therapy with undetectable viral load for 6 months. Patients with HIV who are receiving effective anti-retroviral therapy and have had an undetectable viral load for at least 6 months are eligible. HIV testing not required in the absence of known history of infection.
* Evidence of chronic hepatitis B virus (HBV) that is detectable on suppressive therapy. Patients with evidence of chronic HBV infection with undetectable HBV viral load on suppressive therapy are eligible. HBV testing not required in the absence of known history of infection.
* History of hepatitis C virus (HCV) infection that has not been cured or that has a detectable viral load. Patients with a history of HCV that has been treated and cured are eligible. Patients with HCV infection who are currently on treatment and have an undetectable HCV viral load are eligible. HCV testing not required in the absence of known history of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-04-02 (Estimated); Study Completion 2029-10-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy of motixafortide on measurable residual disease (MRD) levels | Day 1 before motixafortide and Day 2 (estimated total time is 2 days)
  The efficacy of motixafortide on MRD levels will be measured as the proportion of patients who have at least one of the following, as measured in peripheral blood, before versus after motixafortide: MRD negative to MRD positive conversion, or the 5% absolute increase in MRD level by flow cytometry, or leukemia defining polymerase-chain reaction (PCR) transcript (For fusion-driven leukemias or NPM1 and FLT3-ITD-mutated leukemias) or 5% increase in the VAF of recurrent leukemia associated gene mutations by next-generation sequencing (NGS).

SECONDARY OUTCOMES:
Proportion of patients changing from negative to positive MRD levels | Day 1 before motixafortide and Day 2 (estimated total time is 2 days)
  The proportion will be calculated by number of patients with negative MRD levels at enrollment who had positive MRD levels measured after treatment compared to total number of patients.
Percentage change in variant allele frequency (VAF) levels by next-generation sequencing (NGS) using error-corrected sequencing (MRD-Seq) | Day 1 before motixafortide and Day 2 (estimated total time is 2 days)
Percentage change in VAF levels by NGS using MRD-Seq between bone marrow and peripheral blood assessments | Day 1 before motixafortide and Day 2 (estimated total time is 2 days)
Percentage change in detectable transcript levels by polymerase chain reaction (PCR) | Day 1 before motixafortide and Day 2 (estimated total time is 2 days)
Relapse-free survival (RFS) | From Day 1 through completion of follow-up (estimated total time is 18 months)
  RFS is defined as the duration of time from the date of MRD testing to disease relapse or death from any cause, whichever occurs first. Patients who are alive without disease relapses at the time of database lock for analysis will be censored at the last follow up date. Relapse is defined in the ELN 2022 criteria as bone marrow blasts ≥ 5% or reappearance of blasts in the blood in at least 2 peripheral blood samples at least one week apart or development of extramedullary disease.
Time to next line of therapy | From Day 1 through completion of follow-up (estimated total time is 18 months)
  Measured as the duration of time between initial MRD testing and next line of therapy.
Overall survival (OS) | From Day 1 through completion of follow-up (estimated total time is 18 months)
  OS is defined as the duration of time from the date of MRD testing to death from any cause. Patients who are alive at the time of database lock for analysis will be censored at the last follow up date.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Urrutia, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual, de-identified data that has been published will be available for other investigators with approval from the study's PI and Sponsor.
Supporting Information: Study Protocol
Time Frame: Data will be shared starting 12 months after publication through 24 months after publication.
Access Criteria: Proposed use of data has been approved by the Princpal Investigator and Sponsor. Data will be shared via direct communication with the PI.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu